CLINICAL TRIAL: NCT06891950
Title: Phase 3B, Double-blind, Randomized Study to Evaluate the Safety and Non-inferiority of the Humoral Immune Response of the Butantan Dengue Vaccine in Participants Aged 60 to 79 Years Compared to Participants Aged 40 to 59 Years
Brief Title: Butantan-DV Vaccine in Elderly Populations (DEN-04-IB)
Acronym: DEN-04-IB
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Collaborators: Fundação Butantan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEN-04-IB
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Dengue
Keywords: dengue vaccine; elderly population
MeSH Terms: conditions — Dengue | interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind (60-79 years old) and open-label (40-59 years), three-arm parallel Phase 3b, multicenter study to evaluate the safety and non-inferiority of the humoral immune response of the Butantan Dengue vaccine (Dengue 1,2,3,4 (attenuated)) in participants aged 60 - 79 years (elderly) compared to participants aged 40 to 59 years (adults), with or without previous dengue and healthy based on clinical examination. The 997 participants will be randomized with a 9:3:1 allocation, so that the largest group (60 - 79 years) will be allocated to receive Dengue 1,2,3,4 (attenuated) in a blinded regimen (n=690), the next group (40-59 years) will be allocated to receive Dengue 1,2,3,4 (attenuated) in an open regimen (n=230) and the last (60-79 years) will be allocated to receive placebo (n=77), respectively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Care Provider, Investigator, Outcomes Assessor); double (elderly participants).
  The clinical care team, the professional responsible for the vaccination and the elderly participant will not know which investigational product will be administered.
  Only the pharmacists responsible for storing, preparing and dispensing the investigational product of the study will have access to the unblinded information (randomization code). The allocation of the study product will be revealed only after the completion of the follow-up of the participants and the closing of the database to ensure the evaluation of the long-term safety of the product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dengue 1,2,3,4 (attenuated) vaccine in a single dose older adult (Experimental): Participants (60-79y) receiving Butantan DV (N=690)
  Interventions: Biological: Dengue 1,2,3,4 (attenuated) vaccine
- Dengue 1,2,3,4 (attenuated) vaccine in a single dose adult (Experimental): Participants (40-59y) receiving Butantan DV (N=230)
  Interventions: Biological: Dengue 1,2,3,4 (attenuated) vaccine
- Placebo (Placebo Comparator): Participants (60-79y) receiving Placebo (N=77)
  Interventions: Biological: Dengue 1,2,3,4 (attenuated) vaccine

INTERVENTIONS:
Biological: Dengue 1,2,3,4 (attenuated) vaccine — Each 0.5 mL dose of the lyophilized formulation of Dengue 1,2,3,4 (attenuated) presents an approximate concentration of 103.0 PFU of each vaccine virus rDEN1Δ30-1545, rDEN2/4Δ30(ME)-1495,7163, rDEN3Δ30/31-7164, rDEN4Δ30-7132,7163,8308.

SUMMARY:
This is a randomized, double-blind (60 -79 years) and open-label (40-59 years), three-arm parallel Phase 3b, multicenter study to evaluate the safety and non-inferiority of the humoral immune response of the Butantan Dengue vaccine (Dengue 1,2,3,4 (attenuated)) in participants aged 60 -79 years (elderly) compared to participants aged 40 to 59 years (adults), with or without previous dengue and healthy based on clinical examination.

DETAILED DESCRIPTION:
The study aims to evaluate the non-inferiority of the immune response induced by the Dengue 1,2,3,4 (attenuated) vaccine in participants aged 60 - 79 years old (elderly) compared to participants aged 40 to 59 years on Day 42 + 7 days after vaccination. The primary analysis will include the immunogenicity cohort (n=460 participants, allocated 1:1). The primary outcome is the proportion of neutralizing antibody seroconversion measured by plaque reduction neutralization test (PRNT50), for each dengue serotype, of participants aged 60 - 79 years (elderly) compared with participants aged 40 to 59 years (adults), with or without previous exposure to dengue, on Day 42 + 7 days after vaccination. The primary safety outcome will be the frequency and intensity of solicited and unsolicited adverse reactions from vaccination to Day 22 post-vaccination among participants aged 60 - 79 years and in participants aged 40 to 59 years, with or without prior exposure to dengue. The study will last one year in order to assess the duration of the immune response and serious adverse events (SAE) and events of special interest (SIAE). Throughout the study period, there will be surveillance of suspected and confirmed cases of dengue, chikungunya fever and Zika virus fever. Therefore, if the null hypothesis is rejected, the immunogenicity and safety results of immunobridging will be used to expand the use of Dengue 1,2,3,4 (attenuated) for the age group of 60 - 79 years old.

ELIGIBILITY:
Inclusion Criteria:

* a. Healthy participants aged between 40 and 79 years at the time of study entry, with or without a history of exposure to dengue fever;

  b. Agree to periodic contact by telephone, electronic means, and home visits and to the research center;

  c. Participants with reproductive potential must be using some effective contraceptive method at screening and continue using it for up to 90 days after the intervention; except in cases where the volunteer declares that she is not at risk of becoming pregnant, either by not engaging in sexual activities or by engaging in them in a non-reproductive manner, up to 90 days after vaccination;

  d. Demonstrate intent to participate in the study, documented by the participant's signature of the informed consent form, as well as the study procedures, including completing the Participant Diaries, blood collection, and being available for scheduled study visits and contacts.

Exclusion Criteria:

* a. For female participants with reproductive potential: pregnancy (confirmed by positive β-hCG test), breastfeeding or manifest intention to have sexual practices with reproductive potential without using a contraceptive method in the 90 days following vaccination;

  b. Planned donation of blood, semen or eggs in the 90 days following vaccination;

  c. Evidence of active uncontrolled neurological, cardiac, pulmonary, hepatic or renal disease according to anamnesis or physical examination, at the discretion of the investigator;

  d. Diseases that compromise the immune system, including: decompensated diabetes mellitus, active neoplasms or history of neoplasms in the last five years (except basal cell carcinoma), congenital or acquired immunodeficiencies (including HIV/AIDS), solid organ transplants (heart, liver, pancreas, lung, kidney) or uncontrolled autoimmune diseases according to anamnesis or physical examination, as well as a history of liver failure, heart failure or terminal chronic kidney disease or dialysis;

  e. Behavioral, cognitive, or psychiatric illness that, in the opinion of the principal investigator or his/her medical representative, affects the potential participant's ability to understand and comply with the requirements of the study protocol;

  f. Any abuse of alcohol or drugs in the last 12 months prior to enrollment in the study that has caused medical, professional, or family problems, as indicated by the clinical history;

  g. History of severe allergic reaction or anaphylaxis to the vaccine or components of the study vaccine;

  h. History of asplenia;

  i. Participation in another clinical trial with administration of an investigational product during the six months prior to enrollment in the study or scheduled participation in another clinical trial in the 12 months following enrollment;

  j. Previous participation in a dengue vaccine evaluation study or previous exposure to dengue vaccine;

  k. Use of immunosuppressive therapies six months prior to enrollment in the study or their scheduled use in the 12 months following enrollment. The following immunosuppressive therapies will be considered: antineoplastic chemotherapy, radiotherapy, immunosuppressants to induce tolerance to transplants, monoclonal antibody therapy for the treatment of rheumatological diseases, among others;

  l.Having received an immunosuppressive dose of corticosteroid in the last three months prior to inclusion in the study or administration of an immunosuppressive dose of corticosteroid for the 12 months following inclusion in the study. The dose of corticosteroid considered immunosuppressive is the equivalent of prednisone at a dose of 20 mg/day, for adults, for 14 days (cumulative dose equivalent to at least 280 mg of prednisone). Continuous use of topical or nasal corticosteroid is not considered immunosuppressive;

  m. Having received blood products (transfusions or immunoglobulins) in the last three months prior to inclusion in the study, or scheduled administration of blood products or immunoglobulin in the 12 months following inclusion in the study;

  n. Fever, suspected or measured, in the 72 hours prior to vaccination or axillary temperature ≥ 37.8°C on the day of vaccination (inclusion may be postponed until the potential participant has been fever-free for 72 hours);

  o. Having received a live attenuated virus vaccine in the last 28 days or an inactivated vaccine in the last 14 days prior to inclusion in the study, or having been immunized within 12 months of inclusion in the study;

  p. Any other condition that, in the opinion of the principal investigator or his/her medical representative, may jeopardize the safety or rights of a potential participant or that prevents him/her from complying with this protocol.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 997 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity Primary | Day 42+7 days post-vaccination.
  Proportion of neutralizing antibody seroconversion measured by PRNT50, for each dengue serotype, of participants aged 60 -79 years compared (elderly) with participants aged 40 to 59 years (adults), with or without previous exposure to dengue, on Day 42 + 7 days after vaccination.
Safety Primary 1. | From vaccination to Day 22 + 3 days post-vaccination.
  Frequency and intensity of vaccine-related solicited (local and systemic) adverse events, from vaccination to Day 22 + 3 days post-vaccination, among participants aged 60 - 79 years and in participants aged 40 to 59 years, with or without previous exposure to dengue.
Safety Primary 2. | From vaccination to Day 22 + 3 days post-vaccination.
  Frequency and intensity of vaccine-related unsolicited adverse events, from vaccination to Day 22 + 3 days post-vaccination, in participants aged 60-79 years and in participants aged 40 to 59 years, with or without previous exposure to dengue.

SECONDARY OUTCOMES:
Immunogenicity Secondary 1. | Day 1, Day 42 + 7 days and Day 364 + 28 days after vaccination.
  GMT of neutralizing antibodies, for each dengue serotype, of participants aged 60-79 years and of participants aged 40 to 59 years, with or without previous exposure to dengue, on Day 1, Day 42 + 7 days and Day 364 + 28 days after vaccination.
Immunogenicity Secondary 2. | Day 42 + 7 days after vaccination.
  GMT ratio of neutralizing antibodies, for each dengue serotype, of participants aged 60-79 years compared with participants aged 40 to 59 years, with or without previous exposure to dengue, on Day 42 + 7 days after vaccination.
Immunogenicity Secondary 3. | Day 364 + 28 days after vaccination.
  GMT ratio of neutralizing antibodies, for each dengue serotype, of participants aged 60-79 years compared with participants aged 40 to 59 years, with or without previous exposure to dengue, on Day 364 + 28 days after vaccination.
Immunogenicity Secondary 4. | Days 42 + 7 days and Day 364 + 28 days after vaccination.
  Valence or seropositivity rate for multiple dengue virus serotypes measured by PRNT50 in participants aged 60-79 years and in participants aged 40 to 59 years, with or without previous exposure to dengue, on Days 42 + 7 days and Day 364 + 28 days after vaccination.
Safety Secondary 1. | From Day 22 + 3 days post-vaccination until the end of study.
  Frequency and intensity of unsolicited adverse reactions, from Day 22 + 3 days post-vaccination until the end of study follow-up, in elderly participants (60-79 years) and adults (40-59 years), with or without previous exposure to dengue.
Safety Secondary 2. | Throughout the study period.
  Frequency, intensity and causality of serious adverse events, in elderly participants (60-79 years) and adults (40-59 years), with or without previous exposure to dengue, throughout the study period.
Safety Secondary 3. | Throughout the study period.
  Frequency, intensity and causality of adverse events of special interest, in elderly participants (60-79 years) and adults (40-59 years), with or without previous exposure to dengue, throughout the study period.
Safety Secondary 4. | Days 1, 6, 9, 12, 22 and 30.
  Frequency of viremia after vaccination at visits on Days 1, 6, 9, 12, 22 and 30 and laboratory abnormalities in a cohort of 56 elderly participants (60-79 years).
Safety Secondary 5. | Day 29 and throughout the study period.
  Frequency of cases of symptomatic vaccine viremia (Day 29) and of virologically confirmed cases of dengue (VCD), chikungunya fever and Zika virus fever in elderly individuals (60-79 years) and adults (40-59 years), throughout the study period.
Safety Secondary 6. | Day 22 + 3 days after vaccination.
  Frequency of laboratory alterations (aspartate aminotransferase, alanine aminotransferase, total bilirubin, creatinine, blood count) grade 2 or higher among elderly (60-79 years) and adults (40-59 years) on Day 22 + 3 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda C Boulos, MD, PhD, Study Director — Instituto Butantan
Locations (5):
- Brazil (5):
  - CWB 02 - Centro Médico São Francisco, Curitiba, Paraná
  - PET 01 - Hospital Escola da Universidade de Pelotas - HEUFPEL, Pelotas, Rio Grande do Sul
  - POA 05 - Núcleo de Pesquisa do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - POA 02 - Associação Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - POA 01 - Centro de Pesquisa: Hospital São Lucas - PUCRS, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] Gubler DJ. Dengue and dengue hemorrhagic fever. Clin Microbiol Rev. 1998 Jul;11(3):480-96. doi: 10.1128/CMR.11.3.480. PMID 9665979
- [Background] Laydon DJ, Dorigatti I, Hinsley WR, Nedjati-Gilani G, Coudeville L, Ferguson NM. Efficacy profile of the CYD-TDV dengue vaccine revealed by Bayesian survival analysis of individual-level phase III data. Elife. 2021 Jul 2;10:e65131. doi: 10.7554/eLife.65131. PMID 34219653
- [Background] Patel SS, Rauscher M, Kudela M, Pang H. Clinical Safety Experience of TAK-003 for Dengue Fever: A New Tetravalent Live Attenuated Vaccine Candidate. Clin Infect Dis. 2023 Feb 8;76(3):e1350-e1359. doi: 10.1093/cid/ciac418. PMID 35639602
- [Background] Blaney JE Jr, Durbin AP, Murphy BR, Whitehead SS. Development of a live attenuated dengue virus vaccine using reverse genetics. Viral Immunol. 2006 Spring;19(1):10-32. doi: 10.1089/vim.2006.19.10. PMID 16553547
- [Background] Kallas EG, Precioso AR, Palacios R, Thome B, Braga PE, Vanni T, Campos LMA, Ferrari L, Mondini G, da Graca Salomao M, da Silva A, Espinola HM, do Prado Santos J, Santos CLS, Timenetsky MDCST, Miraglia JL, Gallina NMF, Weiskopf D, Sette A, Goulart R, Salles RT, Maestri A, Sallum AME, Farhat SCL, Sakita NK, Ferreira JCOA, Silveira CGT, Costa PR, Raw I, Whitehead SS, Durbin AP, Kalil J. Safety and immunogenicity of the tetravalent, live-attenuated dengue vaccine Butantan-DV in adults in Brazil: a two-step, double-blind, randomised placebo-controlled phase 2 trial. Lancet Infect Dis. 2020 Jul;20(7):839-850. doi: 10.1016/S1473-3099(20)30023-2. Epub 2020 Mar 24. PMID 32220283
- [Background] Kallas EG, Cintra MAT, Moreira JA, Patino EG, Braga PE, Tenorio JCV, Infante V, Palacios R, de Lacerda MVG, Batista Pereira D, da Fonseca AJ, Gurgel RQ, Coelho IC, Fontes CJF, Marques ETA, Romero GAS, Teixeira MM, Siqueira AM, Barral AMP, Boaventura VS, Ramos F, Elias Junior E, Cassio de Moraes J, Covas DT, Kalil J, Precioso AR, Whitehead SS, Esteves-Jaramillo A, Shekar T, Lee JJ, Macey J, Kelner SG, Coller BG, Boulos FC, Nogueira ML. Live, Attenuated, Tetravalent Butantan-Dengue Vaccine in Children and Adults. N Engl J Med. 2024 Feb 1;390(5):397-408. doi: 10.1056/NEJMoa2301790. PMID 38294972
- [Background] Chiaravalloti-Neto F, da Silva RA, Zini N, da Silva GCD, da Silva NS, Parra MCP, Dibo MR, Estofolete CF, Favaro EA, Dutra KR, Mota MTO, Guimaraes GF, Terzian ACB, Blangiardo M, Nogueira ML. Seroprevalence for dengue virus in a hyperendemic area and associated socioeconomic and demographic factors using a cross-sectional design and a geostatistical approach, state of Sao Paulo, Brazil. BMC Infect Dis. 2019 May 20;19(1):441. doi: 10.1186/s12879-019-4074-4. PMID 31109295
- [Background] Schneider M, Narciso-Abraham M, Hadl S, McMahon R, Toepfer S, Fuchs U, Hochreiter R, Bitzer A, Kosulin K, Larcher-Senn J, Mader R, Dubischar K, Zoihsl O, Jaramillo JC, Eder-Lingelbach S, Buerger V, Wressnigg N. Safety and immunogenicity of a single-shot live-attenuated chikungunya vaccine: a double-blind, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 24;401(10394):2138-2147. doi: 10.1016/S0140-6736(23)00641-4. Epub 2023 Jun 12. PMID 37321235
- [Background] Casey RM, Harris JB, Ahuka-Mundeke S, Dixon MG, Kizito GM, Nsele PM, Umutesi G, Laven J, Kosoy O, Paluku G, Gueye AS, Hyde TB, Ewetola R, Sheria GKM, Muyembe-Tamfum JJ, Staples JE. Immunogenicity of Fractional-Dose Vaccine during a Yellow Fever Outbreak - Final Report. N Engl J Med. 2019 Aug 1;381(5):444-454. doi: 10.1056/NEJMoa1710430. Epub 2018 Feb 14. PMID 29443626
- [Background] Hou Y, Chen M, Bian Y, Hu Y, Chuan J, Zhong L, Zhu Y, Tong R. Insights into vaccines for elderly individuals: from the impacts of immunosenescence to delivery strategies. NPJ Vaccines. 2024 Apr 10;9(1):77. doi: 10.1038/s41541-024-00874-4. PMID 38600250
- [Background] Weinberg A, Lazar AA, Zerbe GO, Hayward AR, Chan IS, Vessey R, Silber JL, MacGregor RR, Chan K, Gershon AA, Levin MJ. Influence of age and nature of primary infection on varicella-zoster virus-specific cell-mediated immune responses. J Infect Dis. 2010 Apr 1;201(7):1024-30. doi: 10.1086/651199. PMID 20170376
- [Background] Levin MJ, Oxman MN, Zhang JH, Johnson GR, Stanley H, Hayward AR, Caulfield MJ, Irwin MR, Smith JG, Clair J, Chan IS, Williams H, Harbecke R, Marchese R, Straus SE, Gershon A, Weinberg A; Veterans Affairs Cooperative Studies Program Shingles Prevention Study Investigators. Varicella-zoster virus-specific immune responses in elderly recipients of a herpes zoster vaccine. J Infect Dis. 2008 Mar 15;197(6):825-35. doi: 10.1086/528696. PMID 18419349
- [Background] Collier DA, Ferreira IATM, Kotagiri P, Datir RP, Lim EY, Touizer E, Meng B, Abdullahi A; CITIID-NIHR BioResource COVID-19 Collaboration; Elmer A, Kingston N, Graves B, Le Gresley E, Caputo D, Bergamaschi L, Smith KGC, Bradley JR, Ceron-Gutierrez L, Cortes-Acevedo P, Barcenas-Morales G, Linterman MA, McCoy LE, Davis C, Thomson E, Lyons PA, McKinney E, Doffinger R, Wills M, Gupta RK. Age-related immune response heterogeneity to SARS-CoV-2 vaccine BNT162b2. Nature. 2021 Aug;596(7872):417-422. doi: 10.1038/s41586-021-03739-1. Epub 2021 Jun 30. PMID 34192737
- [Background] Hanley JA, Lippman-Hand A. If nothing goes wrong, is everything all right? Interpreting zero numerators. JAMA. 1983 Apr 1;249(13):1743-5. No abstract available. PMID 6827763
- [Background] Musso D, Ko AI, Baud D. Zika Virus Infection - After the Pandemic. N Engl J Med. 2019 Oct 10;381(15):1444-1457. doi: 10.1056/NEJMra1808246. No abstract available. PMID 31597021
- [Background] Wang WW, Mehrotra DV, Chan IS, Heyse JF. Statistical considerations for noninferiority/equivalence trials in vaccine development. J Biopharm Stat. 2006;16(4):429-41. doi: 10.1080/10543400600719251. PMID 16892905
- [Background] Donken R, de Melker HE, Rots NY, Berbers G, Knol MJ. Comparing vaccines: a systematic review of the use of the non-inferiority margin in vaccine trials. Vaccine. 2015 Mar 17;33(12):1426-32. doi: 10.1016/j.vaccine.2015.01.072. Epub 2015 Feb 7. PMID 25659273
- [Background] Tricou V, Winkle PJ, Tharenos LM, Rauscher M, Escudero I, Hoffman E, LeFevre I, Borkowski A, Wallace D. Consistency of immunogenicity in three consecutive lots of a tetravalent dengue vaccine candidate (TAK-003): A randomized placebo-controlled trial in US adults. Vaccine. 2023 Nov 13;41(47):6999-7006. doi: 10.1016/j.vaccine.2023.09.049. Epub 2023 Oct 24. PMID 37884415
- [Background] Torresi J, Heron LG, Qiao M, Marjason J, Chambonneau L, Bouckenooghe A, Boaz M, van der Vliet D, Wallace D, Hutagalung Y, Nissen MD, Richmond PC. Lot-to-lot consistency of a tetravalent dengue vaccine in healthy adults in Australia: a randomised study. Vaccine. 2015 Sep 22;33(39):5127-34. doi: 10.1016/j.vaccine.2015.08.008. Epub 2015 Aug 13. PMID 26279339
- [Background] LeFevre I, Bravo L, Folschweiller N, Medina EL, Moreira ED Jr, Nordio F, Sharma M, Tharenos LM, Tricou V, Watanaveeradej V, Winkle PJ, Biswal S. Bridging the immunogenicity of a tetravalent dengue vaccine (TAK-003) from children and adolescents to adults. NPJ Vaccines. 2023 May 25;8(1):75. doi: 10.1038/s41541-023-00670-6. PMID 37230978
- [Background] Miettinen O, Nurminen M. Comparative analysis of two rates. Stat Med. 1985 Apr-Jun;4(2):213-26. doi: 10.1002/sim.4780040211. PMID 4023479
- [Result] Nogueira ML, Cintra MAT, Moreira JA, Patino EG, Braga PE, Tenorio JCV, de Oliveira Alves LB, Infante V, Silveira DHR, de Lacerda MVG, Pereira DB, da Fonseca AJ, Gurgel RQ, Coelho IC, Fontes CJF, Marques ETA, Romero GAS, Teixeira MM, Siqueira AM, Boaventura VS, Ramos F, Junior EE, de Moraes JC, Whitehead SS, Esteves-Jaramillo A, Shekar T, Lee JJ, Macey J, Kelner SG, Coller BG, Boulos FC, Kallas EG; Phase 3 Butantan-DV Working Group. Efficacy and safety of Butantan-DV in participants aged 2-59 years through an extended follow-up: results from a double-blind, randomised, placebo-controlled, phase 3, multicentre trial in Brazil. Lancet Infect Dis. 2024 Nov;24(11):1234-1244. doi: 10.1016/S1473-3099(24)00376-1. Epub 2024 Aug 5. PMID 39116904